CLINICAL TRIAL: NCT06626997
Title: Nutritional Intervention Study to Evaluate the Effect of a Symbiotic Drink on the Microbiota and Different Nutritional Markers in Healthy Volunteers
Brief Title: Effect of a Symbiotic Drink on the Microbiota
Acronym: KOMFIBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IMDEA Food (Other)
Responsible Party: Principal Investigator, María Isabel Espinosa, Principal Investigator, IMDEA Food
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IMD: PI-060
Record Dates: First submitted 2024-09-30; First posted 2024-10-04 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: Kombucha; Microbiota
MeSH Terms: interventions — Kombucha Tea

STUDY DESIGN:
Intervention Model Description: Prospective, parallel, randomized 6-week nutritional intervention study.
Who Masked: Participant, Investigator
Masking Description: The study will be masked by using identical packaging for both the study group and the control group (placebo), which participants will consume at home or at their mealtimes during the 6 weeks of the intervention.
  The researchers themselves will administer the product (with identical external appearance for both groups) individually to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study Group (Experimental): Participants will consume a 250cl bottle of soluble fibre-enriched kombucha mid-morning or mid-afternoon, avoiding consumption after eating. The drink will be included in a healthy eating plan. They will be advised to continue their usual physical activity during the 6 weeks of the study.
  Interventions: Dietary Supplement: Kombucha tea
- Control Group (Placebo Comparator): Participants will consume one 250cl bottle of a similar unfermented and unfortified beverage mid-morning or mid-afternoon, avoiding consumption after eating. The beverage will be included in a healthy eating plan. Participants will be advised to continue their usual physical activity for the 6 weeks of the study.
  Interventions: Dietary Supplement: Kombucha tea

INTERVENTIONS:
Dietary Supplement: Kombucha tea — During Visit 1 (week 0), a fasting blood test must be performed at the IMDEA Alimentación facilities to obtain different markers: blood lipids, blood glucose, etc. Approximately 20 mL will be extracted (for comparison, keep in mind that a donation requires 450 mL). The blood sample will be extracted by qualified nursing staff from the UNILABS Laboratory. The blood tests based on the security and privacy requirements for handling samples will be carried out by the same laboratory.
  You will also be asked to provide the stool sample that you must have collected at home prior to attending that visit with the material provided at the screening visit (V0) and at the intermediate visit (V2).

SUMMARY:
This study is expected to involve 60 volunteers who will be recruited by IMDEA-Alimentación and randomly assigned between a study group (which will consume the fermented drink) and a control group, which will consume a drink with similar characteristics, but without the presence of bioactive components.

DETAILED DESCRIPTION:
At the beginning of the trial, you will have an interview (screening visit) with a dietician-nutritionist who will explain the entire procedure to you and answer any questions you may have about it. If it is confirmed that you meet the criteria to participate in the study, after your assent and informed consent have been obtained, you will be able to do so. At the first visit, you will be assigned a code by a random method (computerized) and neither you nor the researcher will know whether you are receiving the enriched product or the traditional one that will be used as a control.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 18 years of age.
* Caucasian ethnicity
* Adequate level of culture and understanding of the clinical study.
* Agree to voluntarily participate in the study and give written informed consent.

Exclusion Criteria:

* Subjects with dementia, mental illness or decreased cognitive function that prevents the study from being carried out.
* Subjects with serious diseases (liver, kidney, immunosuppressed, etc.).
* BMI ≥ 30 kg/m2, pregnant or breastfeeding women.
* Presence of immunological pathologies, gallstones, gastric ulcer or coagulation problems.
* Presence of any other specific pathology that contraindicates the intake of dietary supplements, specifically inulin and probiotics (diverticulitis, etc.).
* Subjects who are undergoing antibiotic treatment or consuming probiotic supplements.
* Subjects who are undergoing pharmacological treatment for weight loss.
* Subjects who refuse to follow the guidelines for healthy eating or the consumption of the study drink in the indicated guidelines.
* Any other exclusion criteria that the principal investigator of the study considers relevant.
* Non-Caucasian ethnicity

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Relative abundance of the gut microbial species | 6 weeks
  Analyze the variations in the relative abundance of the microbial species present, including taxonomic identification, diversity analysis, and phylogenetic composition.

CONTACTS AND LOCATIONS:
Locations (1):
- Imdea Food, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Arce-Lopez B, Bazan GX, Molina S, Crespo MC, Garcia-Beccaria M, Cruz-Gil S, Fernandez-Diaz CM, Ramirez de Molina A, Ramos-Ruiz R, Espinosa-Salinas MI. Effect of fiber-modified kombucha tea on gut microbiota in healthy population: A randomized controlled trial (RCT). Curr Res Food Sci. 2025 Jun 26;11:101130. doi: 10.1016/j.crfs.2025.101130. eCollection 2025. PMID 40689297